CLINICAL TRIAL: NCT04854317
Title: Endoscopic Gastroplasty for Treatment of Obesity: a Single Centre, Randomized Trial
Brief Title: Bariatric Endoscopy for Treatment of Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mater Olbia Hospital (Other)
Responsible Party: Principal Investigator, Salvatore F. Vadalà di Prampero, Principal Investigator, Mater Olbia Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0001501/12/05/2020
Record Dates: First submitted 2021-04-01; First posted 2021-04-22 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Obesity
Keywords: Weight; Obese; Endoscopic Sleeve Gastroplasty; Endoluminal Vertical Gastroplasty; Primary Obesity Surgical Endolumenal 2
MeSH Terms: conditions — Obesity; Body Weight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients undergoing Endoscopic Sleeve Gastroplasty (Active Comparator): Obese patients with I, II, and III grade of obesity (BMI 30-44.99 kg/m2) and previous failed attempts of diet.
  Interventions: Procedure: Endoscopic gastroplasty
- Patients undergoing Endoluminal Vertical Gastroplasty (Active Comparator): Obese patients with I, II, and III grade of obesity (BMI 30-44.99 kg/m2) and previous failed attempts of diet.
  Interventions: Procedure: Endoscopic gastroplasty
- Patients undergoing Primary Obesity Surgical Endolumenal 2 (Active Comparator): Obese patients with I, II, and III grade of obesity (BMI 30-44.99 kg/m2) and previous failed attempts of diet.
  Interventions: Procedure: Endoscopic gastroplasty

INTERVENTIONS:
Procedure: Endoscopic gastroplasty — Endoscopic Gastroplasty
  Other Names: Apollo Overstitch Sx; Endomina; POSE2

SUMMARY:
A single-center, randomized trial will be conducted in order to compare three Endoscopic Gastroplasty (EG) techniques in obese patients (BMI 30-44.99 kg/m2) at Gastroenterology and Gastrointestinal Endoscopy Unit, Mater Olbia Hospital, Qatar Foundation Endowment & Gemelli Foundation, Italy in period June 2020 - August 2024, with the aim to compare the efficacy and safety of these procedures.

DETAILED DESCRIPTION:
BACKROUND Obesity has reached epidemic proportions in the world affecting nowadays, along with overweight, over a third of the world's population. It is a chronic multifactorial illness that can lead to potentially life threatening diseases (such as metabolic disorders, cardiovascular disease, stroke, liver disease, and cancer) that can be prevented and improved by weight loss.

A widely accepted option for the treatment of obesity is the endoscopic approach by many different techniques, ranging from the placement of an intragastric balloon (IGB) to the EG, that are nowadays available in the clinical practice as three techniques: Endoscopic Sleeve Gastroplasty (ESG) with Overstitch Endoscopic Suturing Device (Apollo Overstitch), Endoluminal Vertical Gastroplasty (EVG) with an endoluminal-suturing device (Endomina), and Primary Obesity Surgery Endolumenal-2 (POSE-2). Basically, Bariatric Endoscopy (BE) has two mechanism of action. The first one consists in reduction of the stomach capacity and the second one is alteration of gastric motility.

The major advantages of BE techniques consist in their lower invasiveness compared to surgery, reversibility, short hospital stay, and cost-effectiveness. For instance, laparoscopic sleeve gastrectomy (LSG) is the most performed bariatric surgery procedure that is effective but is associated with important adverse events as bleeding from the staple line that can occur in up to 5% of the procedures, gastric leak and persistent fistulas that can occur in up to 8% the LSG.

The weight reduction is conditioned by patient gastric capacity and treatment duration but also the change in the attitude of the patient towards food and physical activity may be fundamental. It is therefore important that the patient is motivated to lose weight and aware of the consequences of his behaviour.

As at the moment many BE techniques are available and most of them are often interchangeable, it could be important to start clarifying if there are any differences among them in terms of their safety and efficacy.

In this study we focused on EG as literature shows more promising results in terms of weight loss compared to IGB.

TYPE OF STUDY Single centre, randomized trial.

OBJECTIVES Primary objective of the study is to detect any difference among the three EG techniques available in the clinical practice, in terms of weight loss over a 18 months period.

TRIAL DESIGN All patients with indication to EG will be revised by an internal multidisciplinary team composed of gastroenterologist, surgeon, dietitian, psychiatrist, radiologist and endocrinologist.

Before each EG procedure, the patients will be subjected to a psychoclinical assessment (a clinical interview along with psychometric tests) to identify psychopathological conditions which may contraindicate the treatment or personality traits that may predict a successfull treatment (Millon Clinical Multiaxial Inventory-III, MCMI-III); during this visit it will be also evaluated the patients' food-related behavior (Eating Problem Checklist EPCL), their binge eating severity (Binge Eating Scale BES), various aspects of body-image perception and body attitudes (Body Uneasiness Test BUT), the eating impulsivity (BIS-11 Barratt Impulsiveness Scale BIS-11), and the patients' quality of life based on a combination of generic and specific instruments (Obesity Related Well-Being questionnaire ORWELL 97), collateral QoL measures (as the Short Form of SF-36 health Survey, SF-12), together with the patients' own intervention; major endocrine disorders will be excluded and an esophagogastroduodenoscopy will be performed in order to exclude also endoscopic contraindications to the endoscopic bariatric procedure.

Before each EG procedure patients also will get their first dietician examination while at hospital. During the first visit, all patients will be subjected to a clinical interview in order to estimate their calories intake, their eating and taste habits and their level of physical activity, then will be collected anthropometric data (height, weight, circumferences) in order to calculate Body Mass Index (BMI), Waist/Hips ratio (WHR) and cardiovascular risk. Furthermore the dietician will identify a goal for each patient in terms of weight loss and physical activity improvement per week, reinforcing successful outcomes and rewarding good behaviors, also through the involvement of patients family members as social support. Just after the endoscopic bariatric procedure patients will be given a two months refeeding protocol, different depending on endoscopic procedure.

Before the preliminary esophagogastroduodenoscopy a blood sample will be collected in order to establish the initial blood asset for each patient.

A liver ultrasound with elastography will be performed in order to evaluate the degree of steatosis. A transit study examination and a barium x-ray will be performed in order to test the motility and the size of the stomach before the endoscopic bariatric procedure.

After informed consent will be obtained, patients will be randomly enrolled to each procedure, according a software released by the GraphPad Software Company.

Each procedure will be performed by two skilled endoscopists in obesity procedures and with an anaesthesiologist support for monitoring and general anesthesia.

The patients will be randomly divided as follows:

* 1/3 patients will be treated with ESG (created by a series of endoluminally placed free-hand, full-thickness, closely spaced sutures through the gastric wall from the pre-pyloric antrum to the gastroesophageal junction by using an endoscopic suturing device called Overstitch. This procedure reduces the entire stomach along the greater curvature, to form an endoscopically created sleeve);
* 1/3 patients will be treated with POSE2 (large, overtube-style platform that has 4 working channels that can accommodate a slim endoscope and 3 specialized instruments to place transmural tissue anchor plications in parts of the gastric body);
* 1/3 patients will be treated with EVG (by using an over-the-scope triangulation platform attached to an endoscope, anterior-to-posterior greater curvature plications are applied).

After the procure the patients will undergo a dietician check at 30±15, 90±30, 180±30, 360±30, 540±30 days of follow-up. Just after the first follow-up patients will be given a new customized food plan. During each dietician check will be collected new anthropometric data and patients will be trained to reduce calories intake, to increase physical activity, to self-monitoring, to slower eating and they will undergo a nutritional education in order to obtain behavior-change intervention. During dietician checks, the patients will be interviewed regarding their quality of life according the Weiner's Bariatric Quality of Life Index , their behavior change about diet and calories intake and will be collected new anthropometric data in order to evaluate the % of total body weight loss (TBWL%), % of excess weight loss (EWL%) and the Δ Body Mass Index (ΔBMI). Dietician checks will be performed by a dietician who is skilled both in dietician support and behavioral therapy for obese patients.

Furthermore during the follow-up patients will also undergo a psychological visits, with the same timing of the dietician checks (at 30±15, 90±30, 180±30, 360±30, 540±30 days of follow-up), in order to evaluate the compliance to the previous given instructions, to reinforce good eating behaviors and, after a psychoclinical reassessment through some of the above mentioned tests, to give a psychological support in case of need.

Patients will undergo also a gastroenterological visit at 30±15, 90±30, 180±30, 360±30, 540±30 days of follow-up to assess any possible adverse event to the procedure or to modify therapy in case of symptoms not well controlled.

A liver ultrasound with elastography, a transit study examination and a barium x-ray will be performed 3 months after the procedure in order to evaluate any change in hepatic steatosis, motility and size of the stomach.

Blood samples will be collected 30±15 90±30, 180±30, 360±30, 540±30 days after each EG in order to evaluate hormonal and microbiota modifications.

PATIENTS One hundred eighty-nine adult patients with obesity eligible for EG will be randomly and consecutively enrolled in one Endoscopy Unit: Mater Olbia Hospital (Olbia, Italy).

SAMPLE SIZE Assuming from the literature that the bariatric endoscopic techniques considered in our protocol have similar results in the short-term period (i.e. 15-20% of % Total Body Weight Loss), while assuming more relevant differences in the long-term period, a total sample size of 159 patients (53 for each group) will be sufficient to detect a difference of means among the 3 groups, considering an effect size of 25%, a power of 80% and a significance level of 5%. However, to compensate for potential drop-out, enrollment could be continued beyond the planned sample size, with patients allocated to available procedures at the time of enrollment.

STATISTICS Sample characteristics will be summarized as mean ± standard deviation (SD) or median and 25°-75° percentiles (IQR) for quantitative variables, and by absolute and relative (percentages) frequencies for qualitative ones. Shapiro-Wilk test will be used to assess normality f data distribution. Relationship between two quantitative variables will be assessed by calculating Pearson or Spearman correlation coefficients. Pearson Chi Square or Fisher exact tests will be used to evaluate differences of qualitative variables. Differences in quantitative variables between groups will be investigated with unpaired t-test or one-way analysis of variance (ANOVA), as appropriate, or non-parametric methods (Mann-Whitney's and Kruskal-Wallis' tests) if assumptions of parametric tests will be not satisfied. For post hoc multiple testing, we will adjust the alpha level by using the Bonferroni correction (i.e. results were considered statistically significant at p<0.05). For all other analyses, a p-value less than 0.05 will be considered statistically significant. SPSS or Jamovi version 2.2.5 (The jamovi project, Newcastle, Australia) software will be used for statistical computation.

INFORMED CONSENT STATEMENT All patients will be required to give informed consent to the study. All clinical data will be obtained after each patient agreed to treatment by written consent.

DATA RETENTION Data will be retained by the Mater Olbia Hospital in the electronic archive provided for each patient during their first admission at Hospital, as it always happens for all patients.

INSURANCE All patients will be covered by the regular insurance provided by the Mater Olbia Hospital for inpatients and outpatients as the same steps are scheduled also for each patient who should undergo an endoscopic bariatric procedure out of this study.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old;
* acceptance of written informed consent to undergo an EG;
* capability to understand and comply with the study protocol;
* obesity: a BMI of 30-34.99 kg/m2 with previous failed attempts at diet and with obesity-related diseases, a BMI of 35-39.99 kg/m2 with previous failed attempts at diet and with or without obesity-related diseases, a BMI of 40-44.99 kg/m2 with previous failed attempts at diet and with or without obesity-related diseases not fit for surgery.

Exclusion Criteria:

* patients who do not give their consent to the enrollment in the study or are incompetent, unconscious or unable to express their consent for any reason;
* patients suffering from any condition which precludes compliance with study instructions;
* patients who underwent previous attempts at surgical or endoscopic bariatric therapy;
* patient has any allergy or other known contraindication or intolerance to the medications used in the study;
* women who are either pregnant or nursing at the time of screening, or are of child-bearing potential and do not practice methods of contraception;
* patient suffers from a life threatening condition.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2020-06-19 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of Total Body Weight Loss (TBWL percent) | at 30±15, 90±30, 180±30, 360±30, 540±30 days after the procedure
  To evaluate the percentage of Total Body Weight Loss after each endoscopic bariatric procedure

SECONDARY OUTCOMES:
Percentage of Excess Weight Loss (EWL percent) | at 30±15, 90±30, 180±30, 360±30, 540±30 days after the procedure
  To evaluate the percentage of Excess Weight Loss after each endoscopic bariatric procedure
Safety in terms of occurrance intra-procedural, post-procedural and late adverse events (AEs). | intra-procedural, up to 14 days and any time after 14 days
  bleeding (YES/NO), perforation (YES/NO), fistula (YES/NO)
Technical success rate | intra-procedural
  percentage of procedures completed without abortion
Pain procedure-related | the day before the procedure, at 12, 24 hours after the procedure
  NRS pain scale (0-10 points, where 0 is no pain and 10 is the worst pain imaginable)
Vomit procedure-related | at 12, 24 hours after the procedure
  PONV vomit scale 0-3 points (0= no vomit, 1=1 episodes per day, 2= 2 episodes per day, 3= 3 or more episodes per day)
Nausea procedure-related | at 12, 24 hours after the procedure
  PONV nausea intensity scale 0-3 points (0= no nausea, 1=sometimes, 2= often or most of the time, 3= all of the time)
Procedure time differences among the procedures used | intra-procedural
  procedure time (minutes)
Quantity of devices and accessories used during the procedures | intra-procedural
  number of suturing systems, needles, threads, sutures and cinchs
Quality of life (QoL) of endoscopic bariatric procedures | before the procedure (when required by the test) and 1,3,6,12,18,24,36 months after the procedure
  BAROS QoL Scale (BAROS questionnaire), EQ-5D test, Sio test, Scl-90 test, EDE-q, BUT test, DERS test
Hepatic steatosis | before the procedure (at baseline) and 3±1 months after the procedure
  quantification of the hepatic steatosis before and after the procedure by elastography
Transit time | before the procedure (at baseline) and 3±1 months after the procedure
  evaluation of the transit time thorough the stomach by a X-ray with barium meal.

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore F. Vadalà di Prampero, MD, PhD, Principal Investigator — Gastroenterology and GI Endoscopy; Milutin Bulajic, MD, PhD, Study Chair — Gastroenterology and GI Endoscopy
Locations (1):
- Mater Olbia Hospital, Olbia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hruby A, Hu FB. The Epidemiology of Obesity: A Big Picture. Pharmacoeconomics. 2015 Jul;33(7):673-89. doi: 10.1007/s40273-014-0243-x. PMID 25471927
- [Background] Kopelman PG. Obesity as a medical problem. Nature. 2000 Apr 6;404(6778):635-43. doi: 10.1038/35007508. PMID 10766250
- [Background] Yasawy MI, Al-Quorain AA, Hussameddin AM, Yasawy ZM, Al-Sulaiman RM. Obesity and gastric balloon. J Family Community Med. 2014 Sep;21(3):196-9. doi: 10.4103/2230-8229.142977. PMID 25374473
- [Background] ASGE Bariatric Endoscopy Task Force; ASGE Technology Committee; Abu Dayyeh BK, Edmundowicz SA, Jonnalagadda S, Kumar N, Larsen M, Sullivan S, Thompson CC, Banerjee S. Endoscopic bariatric therapies. Gastrointest Endosc. 2015 May;81(5):1073-86. doi: 10.1016/j.gie.2015.02.023. Epub 2015 Mar 28. No abstract available. PMID 25828245
- [Background] ASGE Bariatric Endoscopy Task Force and ASGE Technology Committee; Abu Dayyeh BK, Kumar N, Edmundowicz SA, Jonnalagadda S, Larsen M, Sullivan S, Thompson CC, Banerjee S. ASGE Bariatric Endoscopy Task Force systematic review and meta-analysis assessing the ASGE PIVI thresholds for adopting endoscopic bariatric therapies. Gastrointest Endosc. 2015 Sep;82(3):425-38.e5. doi: 10.1016/j.gie.2015.03.1964. Epub 2015 Jul 29. PMID 26232362
- [Background] Gomez V, Woodman G, Abu Dayyeh BK. Delayed gastric emptying as a proposed mechanism of action during intragastric balloon therapy: Results of a prospective study. Obesity (Silver Spring). 2016 Sep;24(9):1849-53. doi: 10.1002/oby.21555. Epub 2016 Jul 28. PMID 27465076
- [Background] Abu Dayyeh BK, Acosta A, Camilleri M, Mundi MS, Rajan E, Topazian MD, Gostout CJ. Endoscopic Sleeve Gastroplasty Alters Gastric Physiology and Induces Loss of Body Weight in Obese Individuals. Clin Gastroenterol Hepatol. 2017 Jan;15(1):37-43.e1. doi: 10.1016/j.cgh.2015.12.030. Epub 2015 Dec 31. PMID 26748219
- [Background] Nielsen AW, Helm MC, Kindel T, Higgins R, Lak K, Helmen ZM, Gould JC. Perioperative bleeding and blood transfusion are major risk factors for venous thromboembolism following bariatric surgery. Surg Endosc. 2018 May;32(5):2488-2495. doi: 10.1007/s00464-017-5951-9. Epub 2017 Nov 3. PMID 29101558
- [Background] Berger ER, Clements RH, Morton JM, Huffman KM, Wolfe BM, Nguyen NT, Ko CY, Hutter MM. The Impact of Different Surgical Techniques on Outcomes in Laparoscopic Sleeve Gastrectomies: The First Report from the Metabolic and Bariatric Surgery Accreditation and Quality Improvement Program (MBSAQIP). Ann Surg. 2016 Sep;264(3):464-73. doi: 10.1097/SLA.0000000000001851. PMID 27433904
- [Background] Inaba CS, Koh CY, Sujatha-Bhaskar S, Silva JP, Chen Y, Nguyen DV, Nguyen NT. One-Year Mortality after Contemporary Laparoscopic Bariatric Surgery: An Analysis of the Bariatric Outcomes Longitudinal Database. J Am Coll Surg. 2018 Jun;226(6):1166-1174. doi: 10.1016/j.jamcollsurg.2018.02.013. Epub 2018 Mar 16. PMID 29551698
- [Background] Ricca V, Mannucci E, Moretti S, Di Bernardo M, Zucchi T, Cabras PL, Rotella CM. Screening for binge eating disorder in obese outpatients. Compr Psychiatry. 2000 Mar-Apr;41(2):111-5. doi: 10.1016/s0010-440x(00)90143-3. PMID 10741889
- [Background] Marano G, Cuzzolaro M, Vetrone G, Garfinkel PE, Temperilli F, Spera G, Dalle Grave R, Calugi S, Marchesini G; QUOVADIS Study Group. Validating the Body Uneasiness Test (BUT) in obese patients. Eat Weight Disord. 2007 Jun;12(2):70-82. doi: 10.1007/BF03327581. PMID 17615491
- [Background] Fossati A, Di Ceglie A, Acquarini E, Barratt ES. Psychometric properties of an Italian version of the Barratt Impulsiveness Scale-11 (BIS-11) in nonclinical subjects. J Clin Psychol. 2001 Jun;57(6):815-28. doi: 10.1002/jclp.1051. PMID 11344467
- [Background] Mannucci E, Ricca V, Barciulli E, Di Bernardo M, Travaglini R, Cabras PL, Rotella CM. Quality of life and overweight: the obesity related well-being (Orwell 97) questionnaire. Addict Behav. 1999 May-Jun;24(3):345-57. doi: 10.1016/s0306-4603(98)00055-0. PMID 10400274
- [Background] Oria HE, Moorehead MK. Bariatric analysis and reporting outcome system (BAROS). Obes Surg. 1998 Oct;8(5):487-99. doi: 10.1381/096089298765554043. PMID 9819079
- [Background] Weiner S, Sauerland S, Fein M, Blanco R, Pomhoff I, Weiner RA. The Bariatric Quality of Life index: a measure of well-being in obesity surgery patients. Obes Surg. 2005 Apr;15(4):538-45. doi: 10.1381/0960892053723439. PMID 15954234
- [Derived] Vadala di Prampero SF, Geraci M, Cosseddu V, Rocchi C, Bazzu P, Simonelli I, Fiorani M, Formichetti J, Manzoni G, Di Maio F, Massidda M, Masia S, Puci M, Sotgiu G, Milano V, Mancini MA, Rinaldi PM, Giustacchini P, Costamagna G, Bulajic M. EFFECTS OF DIFFERENT TECHNIQUES OF ENDOSCOPIC GASTROPLASTY ON WEIGHT LOSS AMONG PATIENTS WITH OBESITY: A RANDOMIZED, SINGLE-CENTER PRAGMATIC TRIAL. Gastrointest Endosc. 2025 Dec 26:S0016-5107(25)02522-2. doi: 10.1016/j.gie.2025.12.271. Online ahead of print. PMID 41456751